CLINICAL TRIAL: NCT01866371
Title: High Resolution Retinal Imaging
Acronym: AOSLO
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 817019; R24EY019861 (NIH)
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Stargardts; Retinitis Pigmentosa; Age-related Macular Degeneration; Choroideremia; Geographic Atrophy
Keywords: Retina; imaging; retinal degeneration
MeSH Terms: conditions — Retinitis Pigmentosa; Macular Degeneration; Choroideremia; Geographic Atrophy; Retinal Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Retinal degeneration: This group will include patients with retinal degeneration and vision abnormalities. The group will participate in retinal imaging procedures including adaptive optics imaging, optical coherence tomography and fundus photography. Vision may be assessed using microperimetry, visual fields, and visual acuity.
  Interventions: Procedure: Retinal imaging
- Normal control: This group will include individuals without retinal degeneration. The group will participate in retinal imaging procedures including adaptive optics imaging, optical coherence tomography and fundus photography. Vision may be assessed using microperimetry, visual fields, and visual acuity.
  Interventions: Procedure: Retinal imaging

INTERVENTIONS:
Procedure: Retinal imaging — Retinal imaging procedures include adaptive optics imaging, optical coherence tomography and fundus photography.

SUMMARY:
Studying the morphology and function of the normal and diseased retina in vivo is needed for advancing the detection, diagnosis, and treatment of retinal disease. This protocol uses an adaptive optics scanning laser ophthalmoscope (AOSLO) to image the normal and diseased retina with individual cellular resolution non-invasively. The primary objective of this study is to obtain and analyze high-resolution images of the retina, in particular by imaging the cone photoreceptor mosaic, the retinal vasculature and other retinal layers. The study design will involve case-control studies, where cases are followed over time. Subjects age 7 and older may be invited to participate. The main research procedure involves retinal imaging with the AOSLO. The primary endpoint is the observation of differences in retinal images between subjects with and without retinal diseases. These changes will be quantified by examining the cell density, size, spacing and regularity of the cone photoreceptor mosaic, as well as examining the differences between other retinal layers.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age 7 years or older.
* Parental/guardian permission (informed consent) and if appropriate, child assent. Child subjects age 7-17 must give assent.
* Reasonable compliance with an imaging protocol as determined by the study personnel.

Exclusion Criteria:

* Individuals that are at risk to acute glaucoma.
* Individuals that are photophobic and experience adverse psychological reactions to flashes of light.
* Ocular opacities, high refractive error, and high frequency of nystagmus as determined by the study team.

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals age 7 and older will be recruited for purposes of this study. Adults must have the capacity to give informed consent. Subjects age 7 to 17 will need parent/guardian consent to participate in the study. Subjects aged 7 to 17 will need to assent to participate in the study. We will recruit subjects with both normal (disease-free) retinas and subjects with retinal degenerations including Leber's Congenital Amaurosis, Stargardt's Dystrophy, retinitis pigmentosa, age-related macular degeneration, Choroideremia, Geographic Atrophy, etc. Subjects will not be excluded based on ethnic or racial background; we expect that enrollment will be split evenly between males and females.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2013-05; Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
high-resolution images of retina | 1 day (initial visit)
  The primary objective of this study is to obtain and analyze high-resolution images of the retina in normal and diseased eyes non-invasively.

SECONDARY OUTCOMES:
Cone mosaic parameters | 1 day (initial visit)
  Imaging the cone photoreceptor mosaic, and analyzing cell density, size, spacing, regularity, and other mosaic parameters in normal retina compared to diseased retina.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica IW Morgan, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Morgan JI, Han G, Klinman E, Maguire WM, Chung DC, Maguire AM, Bennett J. High-resolution adaptive optics retinal imaging of cellular structure in choroideremia. Invest Ophthalmol Vis Sci. 2014 Sep 4;55(10):6381-97. doi: 10.1167/iovs.13-13454. PMID 25190651